CLINICAL TRIAL: NCT01423188
Title: Phase IIb Multi-center, Double-blind, Randomized, Parallel Group, Placebo Controlled Clinical Trial for the Assessment of Lipid Trends and Safety of RVX000222 in Statin Treated Subjects With Low Baseline HDL-C Concentrations
Brief Title: The Study of Quantitative Serial Trends in Lipids With ApolpoproteinA-I Stimulation
Acronym: SUSTAIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Resverlogix Corp (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RVX222-CS-008
Record Dates: First submitted 2011-08-22; First posted 2011-08-25 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: Coronary Artery Disease; Dyslipidemia
Keywords: ApolipoproteinA1; HDL-C; Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Dyslipidemias; Atherosclerosis | interventions — apabetalone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RVX000222, 200 mg daily (Experimental)
  Interventions: Drug: RVX000222
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo RVX000222

INTERVENTIONS:
Drug: RVX000222 — capsule, 200 mg, administer with food, 100 mg twice daily 10-12 hrs apart, 24 weeks
  Arms: RVX000222, 200 mg daily
Drug: Placebo RVX000222 — capsule, administer with food, twice daily 10-12 hrs apart, 24 weeks
  Arms: Placebo

SUMMARY:
This study is designed to provide an assessment of the change in baseline lipid parameters with RVX000222 after 12 weeks and 24 weeks of treatment when given in addition to optimized statin background therapy in subjects with low baseline HDL-C.

DETAILED DESCRIPTION:
One-third of the US population, almost 80 million adults, have cardiovascular disease and mortality associated with heart disease still remains as a leading cause of death around the world. The major risk factors for cardiovascular disease associated with atherosclerosis is dyslipidemia, characterized by high levels of low density lipoprotein (LDL) and/or low levels of high density lipoprotein (HDL). The widespread use of statins in patients at risk for cardiovascular disease has led to lower LDL levels but has had little effect on HDL levels. HDL has a well established role in atherosclerosis and cardiovascular disease protection. HDL mediates the removal of cholesterol from the atherosclerotic plaques for elimination from the body. The major component of HDL consists of apolipoprotein A-I (ApoA I). Recent intervention studies with synthetic HDL particles and recombinant ApoA-I have shown that HDL has the capacity to reverse coronary atherosclerosis. Increasing ApoA-I is likely to have a favorable effect on atherosclerotic plaque stability and size and on cardiovascular diseases. RVX000222 is a member of a novel class of small molecules that are candidates for the treatment of dyslipidemia by increasing plasma levels of HDL through increased ApoA-I transcription.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patient's ≥ 18 years of age with or without documented coronary artery disease
2. Women of child-bearing potential, that is, women not surgically sterilized and between menarche and 1 year post menopause, must test negative for pregnancy at the time of enrollment based on a serum pregnancy test and agree to use a reliable method of birth control (for example, use of oral contraceptives or levonorgestrel); or a reliable barrier method of birth control (diaphragms with contraceptive jelly; cervical caps with contraceptive jelly; condoms with contraceptive foam; intrauterine devices; partner with vasectomy; or abstinence) during the study and for one month following the last dose of study drug.
3. HDL-C requirements. Current (Local lab within 60 days or central lab results prior to Visit 1): HDL-C of ≤45 mg/dL (1.17 mmol/L) for females, and HDL-C of ≤40 mg/dL (1.04 mmol/L) for males
4. Taking statin therapy for at least 30 days prior to screening (Visit 1), and in the investigators opinion, an unlikely need for statin dose adjustment during the course of the study.
5. In the opinion of the investigator patients currently on statin therapy other than atorvastatin (10mg, 20mg or 40mg) or rosuvastatin (5mg, 10mg or 20 mg) can be switched to rosuvastatin (5mg, 10mg or 20mg) at Visit 1.

Exclusion Criteria:

1. Clinically significant heart disease which will require coronary bypass, PCI, cardiac transplantation, surgical repair and/or replacement during the course of the study.
2. Coronary artery bypass graft (CABG) procedure within the past 90 days.
3. Previous or current diagnosis of severe heart failure (NYHA Class III-IV) or a documented left ventricular ejection fraction (LVEF) of <25% as determined by contrast left ventriculography, radionuclide ventriculography or echocardiography the absence of an LVEF measurement in a patient without a previous or current diagnosis of heart failure does not prohibit entry into the study.
4. Patients with evidence of cardiac electrophysiologic instability including a history of uncontrolled ventricular arrhythmias, uncontrolled atrial fibrillation/flutter or uncontrolled supraventricular tachycardias with a ventricular response heart rate of >100 beats per minute at rest within 4 weeks prior to Visit 1.
5. Evidence of renal impairment as determined by any one of the following:

   1. serum creatinine >1.5 mg/dL (>133 micromol/L) at screening Visit 1
   2. a history of dialysis
   3. a history of nephritic syndrome
6. Have hypertension that is uncontrolled defined as 2 consecutive measurements of sitting blood pressure of systolic >160 mm Hg or diastolic >95 mm Hg at Visit 1.
7. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive beta-hCG laboratory test (≥5 mIU/mL).
8. Current or recent (within 12 month prior to Visit 1) treatment with immunosuppressants (eg, Cyclosporine).
9. Triglycerides >400 mg/dL at screening Visit 1.
10. Atorvastatin >40 mg daily
11. Rosuvastatin >20 mg daily
12. Use of fibrates any dose or niacin/nicotinic acid 250 mg or more within 90 days prior to Visit 1.
13. Any medical or surgical condition which might significantly alter the absorption, distribution, metabolism or excretion of medication including, but not limited to any of the following: cholecystitis, Crohn's disease, ulcerative colitis, or any gastric bypass alteration.
14. Evidence of hepatic disease as determined by any one of the following:

    * ALT, AST or GGT values >ULN by central lab at screening, Visit 1
    * a history of hepatic encephalopathy,
    * history of Hepatitis B, C or E,
    * a history of esophageal varices, or
    * a history of portocaval shunt.
15. A total bilirubin that is >ULN by central lab at screening, Visit 1.
16. History of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin.
17. History or evidence of drug or alcohol abuse within the last 12 months.
18. Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study.
19. Use of other investigational drugs and devices at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer.
20. History of noncompliance to medical regimens or unwillingness to comply with the study protocol.
21. Any condition that in the opinion of the investigator would confound the evaluation and interpretation of efficacy and/or safety data.
22. Persons directly involved in the execution of this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The percent change in HDL-C from baseline to 24 weeks for RVX000222 200 mg daily compared to placebo | 24 weeks
  To determine whether treatment with RVX000222 produces an increase in HDL-C at 24 weeks compared to placebo.

SECONDARY OUTCOMES:
Within treatment group percent change in HDL-C from baseline to 24 weeks for RVX000222 and placebo groups. | 24 weeks
  To evaluate changes in other lipids such as HDL-C, LDL-C, non-HDL-C, apoB, TG and HDL subclasses over time within and between treatment groups.
The percent change in plasma apoA-I from baseline to 4 weeks, 12 weeks and 24 weeks for RVX000222 compared to placebo (within and between treatment groups). | 4, 12 and 24 weeks
  To evaluate changes in plasma levels of apoA-I over time within and between treatment groups.
The percent change in LDL-C, non-HDL-C, apoB, TG and HDL subclasses from baseline to 4 weeks, 12 weeks and 24 weeks for RVX000222 compared to placebo (within and between treatment groups) | 4, 12 and 24 weeks
  To evaluate changes in other lipids such as HDL-C, LDL-C, non-HDL-C, apoB, TG and HDL subclasses over time within and between treatment groups.
Incidence of adverse events by treatment group | Participants will be followed for the duration of the study: 30 weeks (2 weeks screening, 24 weeks active treatment, 4 week follow-up)
  To evaluate the safety and tolerability of RVX000222.
The percent change in HDL-C from baseline to 4 weeks and 12 weeks for RVX000222 compared to placebo (within and between treatment groups) | 4, 12 weeks
  To evaluate changes in other lipids such as HDL-C, LDL-C, non-HDL-C, apoB, TG and HDL subclasses over time within and between treatment groups.
The percent change in hsCRP from baseline to 12 weeks and 24 weeks for RVX000222 compared to placebo (within and between treatment groups). | 12, 24 weeks
  To evaluate changes in hs-CRP over time within and between treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Nicholls, MBBS, PhD, Principal Investigator — The Cleveland Clinic
Locations (24):
- South Africa (24):
  - East Burger Street, Bloemfontein
  - Westdene, Bloemfontein
  - Goodwood, Cape Town
  - Kraaifontein, Cape Town
  - Pinelands, Cape Town
  - Chatsworth, Durban
  - KwaKhangela, Durban
  - Merebank, Durban
  - Sydenham, Durban
  - Tongaat, Durban
  - Umhlanga, Durban
  - Lenasia, Johannesburg
  - Halfway House, Midrand
  - Die Wilgers, Pretoria
  - Eloffsdal, Pretoria
  - Kuils River, Western Cape
  - Parow, Western Cape
  - Somerset West, Western Cape
  - Stellenbosch, Western Cape
  - Worcester, Western Cape
  - Bloemfontein
  - Cape Town
  - Johannesburg
  - Western Cape

REFERENCES:
- [Derived] Nicholls SJ, Gordon A, Johannson J, Ballantyne CM, Barter PJ, Brewer HB, Kastelein JJ, Wong NC, Borgman MR, Nissen SE. ApoA-I induction as a potential cardioprotective strategy: rationale for the SUSTAIN and ASSURE studies. Cardiovasc Drugs Ther. 2012 Apr;26(2):181-7. doi: 10.1007/s10557-012-6373-5. PMID 22349989